CLINICAL TRIAL: NCT02525926
Title: Pulmonary Artery Denervation for Treatment of Pulmonary Arterial Hypertension
Acronym: DENERV'AP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Refusal of CPP to extend the period of inclusion
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: Assistance Publique Hopitaux De Marseille (Other); University Hospital, Toulouse (Other); University Hospital, Grenoble (Other); Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-APN-02
Record Dates: First submitted 2015-07-03; First posted 2015-08-18 (Estimated); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Denervation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- denervation (Experimental)
  Interventions: Procedure: denervation
- control group (Sham Comparator)
  Interventions: Procedure: sham procedure

INTERVENTIONS:
Procedure: denervation — The examination proceeds under rigorous aseptic technique. Femoral, jugular or brachial venous access will be performed. A flexible catheter is first introduced across a 7-Fr venous introducer, and passed through the right heart chambers toward the origin of the pulmonary arteries. The pressures in the right heart chambers and the pulmonary artery will be measured. At the end of the examination, the catheter is removed, a dressing is applied and the venous puncture is compressed by hand.
  Arms: denervation
Procedure: sham procedure — Right heart catheterism is mandatory in PAH patients care (for diagnosis and during follow-up) and will serve as a " sham " procedure. A usually performed and after a venous punction, cardiac outpout and pulmonary artery pressures will be recorded.
  Acoustically isolated headphones will be given to patients during the procedure in order to assure simple-blind during the study.
  Arms: control group

SUMMARY:
Pulmonary hypertension is a rare condition that leads to right ventricular dysfunction and premature death. Only modest improvements of outcomes have been observed with the current available advanced specific drug therapy. Pulmonary hypertension advanced therapy is also expensive and leads to frequent adverse effects, sometimes serious. Results from a pilot study, the first-in-man experience of pulmonary artery denervation, demonstrated a clinical improvement in 13 patients with severe pulmonary hypertension despite optimal medical management. However this single non-randomized study requires confirmation.

The investigators propose a prospective multi-center, randomized, single-blinded trial. Its main objective will be to assess, in patients with uncontrolled pulmonary hypertension despite optimal medical management, the efficacy of pulmonary artery denervation in reducing mean pulmonary artery pressure (mPAP) at six months, compared to continued medical treatment following a simulated (sham) procedure.

The principal evaluation criteria will be the mPAP change (in mm Hg) as measured by right heart catheterization.

The study will run for 18 months and it will be necessary to recruit 50 patients.

All adult patients (with the exception of pregnant women and individuals unable to receive an appropriate information and to give their free and informed consent) with uncontrolled pulmonary arterial hypertension despite optimal medical management will be invited to participate, in the absence of any exclusion criteria.

The investigators will also measure changes in clinical, biological, echocardiographic and hemodynamic prognostic markers in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pulmonary artery hypertension (group 1 of the Nice classification of pulmonary hypertension)

  * Aged over 18 years old
  * NYHA class III or IV
  * Not controlled by optimal medical management as defined by:

    * dual therapy including a prostacyclin.
    * or dual therapy including an endothelin receptor antagonist and a
  * 5-phosphodiesterase inhibitors, in patients with contra-indication of prostacyclin, poor tolerance to this treatment, prostacyclin derivative treatment failure or patient refusal.
  * Valid status in the social security system
  * Signed informed consent

Exclusion Criteria:

* Patient eligible for pulmonary transplantation
* Pregnancy or breastfeeding
* Adults of the age of majority subject to guardianship court order or deprived of liberty
* Patient with history of radio frequency procedure
* Known heparin allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-02-04 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Mean pulmonary artery pressure (in mmHg) measured during right heart catheterization | at 6 month

SECONDARY OUTCOMES:
Mean pulmonary artery pressure (in mmHg) from the initial procedure | at 3 month
Pulmonary vascular resistance (in Wood units) measured during right cardiac catheterization. | at 6 month
Clinical parameters: NYHA class | at 6 month
Clinical parameters: Borg dyspnea rating scale | at 6 month
Clinical parameters: 6-minute walk test (distance walked in meters), | at 6 month
Clinical parameters: oxygen dependence (quantity of oxygen in L/min), | at 6 month
Clinical parameters: ECG with supra ventricular arrhythmia. | at 6 month
Biological parameters: levels of Brain Natriuretic Peptide (pg/ml) in non-fasting morning samples. | at 6 month
Biological parameters: levels of troponin Ic (ng/ml) in non-fasting morning samples. | at 6 month
Echocardiographic parameters of right ventricular function | at 6 month
  1. Right ventricular diameter at admission (mm) in 4-chamber view
  2. Right ventricular systolic function: tricuspid annular plane systolic excursion (TAPSE) (mm), peak S-wave velocity at the lateral tricuspid ring (cm/s), Right ventricular fractional area change (%), acceleration (m/s2) and peak isovolumic contraction (cm/s), pulmonary systolic time velocity integral (cm), longitudinal deformation of right ventricular free wall using speckle-tracking imaging (%)
  3. Right ventricular adaptation: right ventricular Tei-index and presence of pericardial effusion
Other hemodynamic parameters obtained by right cardiac catheterization | at 6 month
  1. Cardiac index/output using thermodilution (L/min/m2)
  2. Right atrial pressure (mmHg)

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CHU de Grenoble, Grenoble
  - AP-HM, Marseille
  - CHU de Nice, Nice
  - AP-HP, Paris
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No